CLINICAL TRIAL: NCT03076203
Title: Phase IB Trial of Radium-223 and Niraparib in Patients With Castrate Resistant Prostate Cancer (NiraRad)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Janssen, LP (Industry); Prostate Cancer Clinical Trials Consortium (Other); Bayer (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16G.085; JT 8649 (Other: JeffTrial Number)
Record Dates: First submitted 2017-02-21; First posted 2017-03-10 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Prostate Carcinoma Metastatic to the Bone; Stage IV Prostate Adenocarcinoma; Hormone-refractory Prostate Cancer
MeSH Terms: interventions — niraparib; radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (niraparib, radium Ra 223 dichloride) (Experimental): Patients receive niraparib orally daily and radium Ra 223 dichloride IV over 1 minute every 4 weeks. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Niraparib; Radiation: Radium Ra 223 Dichloride

INTERVENTIONS:
Drug: Niraparib — Given orally
  Other Names: MK4827; MK-4827
Radiation: Radium Ra 223 Dichloride — Given intravenously
  Other Names: BAY 88-8223; Radium 223 Dichloride; RADIUM CHLORIDE RA-223; Xofigo

SUMMARY:
This phase Ib trial studies the side effects and best dose of niraparib when given together with radium Ra223 dichloride in treating subjects with prostate cancer that keeps growing even when the amount of testosterone in the body is reduced to very low levels and has spread from the primary site to the bone. Radium Ra 223 dichloride, acts like calcium to target cancer in the bones and may deliver radiation directly to the bone tumors, limiting damage to the surrounding normal tissue. Niraparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving radium Ra 223 dichloride and niraparib may work better in treating subjects with hormone-resistant prostate cancer metastatic to the bone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine a safe dose of niraparib when combined with radium Ra 223 dichloride (radium-223) in patients with metastatic castrate-resistant prostate cancer (mCRPC) that have and have not received prior chemotherapy.

SECONDARY OBJECTIVES:

I. To determine the proportion of subjects with 50% prostate-specific antigen (PSA) reduction from baseline in men treated with niraparib and radium 223.

II. To determine the radiographic PFS (rPFS) at 6 months in men treated with niraparib and radium 223.

III. To determine the proportion of subjects that have circulating tumor cell (CTC) conversion (>= 5 to < 5/7.5ml) confirmed in a second assessment > 4 weeks later in men treated with niraparib and radium 223.

IV. To determine the overall progression-free survival in men treated with niraparib and radium 223.

V. To determine the time to total-ALP (alkaline phosphatase) progression defined in subjects with no total-ALP decline from baseline as >= 25% increase from the baseline value, at least 12 weeks from baseline.

VI. To determine the time to total-ALP (alkaline phosphatase) progression defined in patient with an initial total-ALP decline from baselines as >= 25% increase from the nadir value, which is confirmed by a second value obtained three or more weeks later.

VII. To determine the total-ALP normalization, defined as the return of total-ALP value to within normal range at 12 weeks in 2 consecutive measurements (at least 2 weeks apart) after that of treatment in subjects who have their ALP above upper limit of normal (ULN) at baseline.

VIII. To determine the long term safety-tolerability of the combination of niraparib and radium 223 in men treated with niraparib and radium 223.

TERTIARY OBJECTIVES:

I. Study of deoxyribonucleic acid (DNA) repair aberrations; whole exome and transcriptome in pre-therapy tumor biopsy samples.

II. Compare changes in bone marrow micro-environment (hematopoietic stem cell [HSC] niche\ C-X-C motif chemokine ligand 12 [CXCL12]/C-X-C motif chemokine receptor 4 [CXCR4] axis) pre and post therapy in up to 10 men treated with niraparib and radium 223.

III. Evaluate the baseline plasma cell-free (cf)-DNA for aberrations in DNA repair genes such as breast cancer (BRCA)1, BRCA2, ataxia telangiectasia mutated (ATM), ataxia-telangiectasia and rad3-related (ATR), partner and localizer of brca2 gene (PALB2) as well as the androgen receptor (AR) gene via next generation sequencing.

IV. Compare gene expression changes in baseline and serial (at end of cycle 1 and 3) whole blood ribonucleic acid (RNA) (collect blood in edetic acid [EDTA] tubes and RNA-later) using Nanostring PanCancer and immunology panel.

V. Evaluate the baseline CTCs for nuclear androgen receptor (AR), phosphorylated (p) nuclear factor kappa-beta (NF-kB), and gamma-H2A histone family member X (H2AX) foci via immunostaining.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
* Bone metastases
* Documented progressive metastatic CRPC based on at least one of the following criteria:

  * PSA progression defined as a miminum of 2 rising PSA levels with a minimum of a 1 week interval and a minimum PSA of 2 ng/mL

    -1.0 ng/mL is the minimal starting PSA value if confirmed rise is the only indication of progression
  * Soft-tissue progression defined as an increase >= 20% in the sum of the longest diameter (LD) of all target lesions based on the smallest sum LD since treatment started or the appearance of one or more new lesions or the appearance of new lesions
  * Documented appearance of new lesions by bone scan
* Agree to undergo a tumor/bone marrow biopsy or submit archival tissue. Note: Tissue sample collected from primary or metastatic site is acceptable on study. Once each stratum begins enrollment at the 300mg dose level, 5 subjects from each stratum will complete a bone marrow biopsy. Due to the dose assignment method used in this study, the 10 subjects requiring a bone marrow biopsy on study will be determined on a case by case basis after consent
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Must have received at least 1 line of AR-targeted therapy or androgen bio-synthesis inhibitor (e.g., abiraterone acetate, enzalutamide, apalutamide) for prostate cancer
* Testosterone =< 50 ng/dL; subjects must continue primary androgen deprivation with an luteinizing hormone-releasing hormone (LHRH) analogue (agonist or antagonist) if they have not undergone orchiectomy
* Subjects on long term (>= 6 months) first generation anti-androgen therapy (e.g. flutamide, bicalutamide, nilutamide) will need to discontinue anti-androgen therapy for 4 weeks (wash out period) and show evidence of disease progression off the anti-androgen; subjects that have been on a first generation anti-androgen 6 months or less will need to discontinue therapy prior to registration (no wash out period required)
* Subjects on second generation anti-androgen therapy (enzalutamide) or androgen bio-synthesis inhibitor (abiraterone acetate) will need to discontinue therapy 2 weeks prior to registration (wash out period)
* Subjects on treatment with chemotherapy or any investigational therapeutic agent will need to discontinue therapy 4 weeks prior to registration (wash out period)
* Absolute neutrophil count (ANC) >= 1,500/uL
* Hemoglobin >= 10 g/dL
* Platelet count >= 150,000/uL
* Creatinine =< 1.5 x the institutional ULN
* Potassium > 3.5 mmol/L (within institutional normal range)
* Total Bilirubin =< 1.5 ULN (unless documented Gilbert's disease)
* Serum glutamic oxaloacetic transaminase (SGOT) aspartate aminotransferase (AST) =< 2.5 x ULN
* Serum glutamate pyruvate transaminase (SGPT) alanine aminotransferase (ALT) =< 2.5 x ULN
* Men must agree to use adequate contraception prior to study entry, for the duration of study participation and for at least 6 months after last radium 223 dose
* Must be able to take oral medication without crushing, dissolving or chewing capsules
* May have received prior radiation therapy or surgery; however, at least 21 days must have elapsed since completion of radiation therapy or surgery and patient must have recovered from all side effects at the time of registration
* Ability to understand and the willingness to sign a written informed consent document that is approved by the local institutional review board

Exclusion Criteria:

* Concurrent treatment with any other investigational therapeutic agents
* More than one prior line of chemotherapy
* More than one prior line of therapy with a second generation anti-androgen (enzalutamide, ARN-509, etc.) or androgen bio-synthesis inhibitor (abiraterone acetate, TAK 700, etc.); patient may have had one second generation anti-androgen or androgen bio-synthesis inhibitor but not both sequentially; subjects that have received combination therapy with second generation anti-androgen plus an androgen bio-synthesis inhibitor would be eligible (e.g., enzalutamide plus abiraterone acetate as one line of therapy on a clinical trial). Note, subjects who have had one line of therapy in a hormone-sensitive setting or one line of therapy in castrate resistant setting are eligible for study.
* Prior isotope therapy with strontium-89, samarium or RAD223
* Subjects with known symptomatic brain metastases
* All herbal, alternative and food supplements (i.e. PC-Spes, saw palmetto, St. John's wort, etc.) must be discontinued before registration; Subjects may continue on a daily multi-vitamin, calcium and vitamin D
* Pre-planned concurrent cytotoxic chemotherapy, surgery, or radiation therapy during protocol treatment; radiation therapy is not permitted while on study
* All hormonal-acting agents (including diethylstilbestrol/DES, aldosterone, and spironolactone) must be discontinued before registration; no washout period will be required for any of these agents
* Initiation of bisphosphonate/denosumab therapy during the study; subjects on stable doses of bisphosphonates or the tumor necrosis factor receptor superfamily member 11a, subfamily L (RANK-L) inhibitor, denosumab, which have been started no less than 4 weeks prior to registration, may continue on this medication
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association class III and IV heart failure), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or concurrent medications that alter cardiac conduction
* Subjects with a "currently active" second malignancy other than non-melanoma skin or superficial urothelial cancers are not eligible; Subjects are not considered to have a "currently active" malignancy if they have completed therapy and are now considered without evidence of disease for 2 years
* Subjects with any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Subjects with known persistent (> 4 weeks) >= grade 2 toxicity from prior cancer therapy
* Subjects with known >= grade 3 hematological toxicity lasting greater than 7 days with the last chemotherapy regimen
* Subjects with chronic conditions associated with non-malignant abnormal bone growth (e.g., Paget's disease of bone)
* Subjects who have used any of the following within 4 weeks prior to registration: blood or platelet transfusions, erythropoietin, and biologic response modifiers such as granulocyte macrophage colony-stimulating factor (GM-CSF) or granulocyte colony-stimulating factor (G-CSF)
* Subjects with baseline QT prolongation > 470 msec
* Subjects receiving concomitant medications that prolong corrected QT interval (QTc)
* Subjects with bulky visceral disease defined as > 4 cm
* Known disorder affecting gastrointestinal absorption
* Subjects with known allergies, hypersensitivity, or intolerance to niraparib or its excipients
* Subjects requiring escalating doses of prednisone or steroids for control of disease at the time of screening. Note: If subjects are receiving prednisone or steroids, they must continue on the same dose they were receiving at the time of screening while being treated on study
* HIV positive subjects with 1 or more of the following:

  * Not receiving highly active antiretroviral therapy
  * A change in antiretroviral therapy within 6 months of the start of screening (except if, after consultation with the sponsor on exclusion criterion 26c. a change is made to avoid a potential drug-drug interaction with the study drug)
  * receiving antiretroviral therapy that may interfere with the study drug (consult the sponsor for review of medication prior to enrollment)
  * CD4 cont <350 at screening
  * An acquired autoimmunodeficiency syndrome-defining opportunistic infection within 6 months of the start of screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of niraparib to combine with radium Ra 223 dichloride based on dose limiting toxicities graded by National Cancer Institute, Common Toxicity Criteria, version 4.0 | 12 weeks
  There will be three dose levels of niraparib combined with standard doses of Radium 223 to be evaluated for safety

CONTACTS AND LOCATIONS:
Overall Officials: William Kelly, DO, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - University of Chicago Medical Center, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/